CLINICAL TRIAL: NCT01458548
Title: Treatment of Patients With Posttransplant Lymphoproliferative Disorder (PTLD) With a Sequential Treatment Consisting of Anti-CD20 Antibody Rituximab and CHOP+GCSF Chemotherapy (Including 1st+2nd Amendment)
Brief Title: Sequential Treatment of CD20-positive Posttransplant Lymphoproliferative Disorder (PTLD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study had an major amendment in 12/2006 introducing risk stratified sequential treatment (RSST). The modified protocol is registered with NCT00590447.
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Ralf Trappe, Head German PTLD Study Group, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTLD-1
Record Dates: First submitted 2011-10-18; First posted 2011-10-25 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Post-transplantation Lymphoproliferative Disorder
Keywords: 1st-line therapy; single agent rituximab; CHOP; PTLD
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rituximab — Rituximab 375 mg/m2 IV on days 1, 8, 15 and 22.
Drug: CHOP — Cyclophosphamide 750 mg/m2 IV, adriamycine 50 mg/m2 IV, vincristine 1.4mg/m2 IV, and prednisone 50mg/m2 PO every 3 weeks at days 50, 72, 94 and 116.

SUMMARY:
Post-transplantation lymphoproliferative disorder (PTLD) develops in one to ten per cent of transplant recipients and can be EBV-associated. To improve long-term efficacy after rituximab monotherapy and to avoid the toxicity of CHOP seen in first-line treatment, the investigators initiated an international multicentre phase II trial to test whether the subsequent application of rituximab and four courses of three-weekly CHOP would improve the outcome of patients with PTLD: PTLD-1, sequential treatment (ST).

ELIGIBILITY:
Inclusion Criteria:

* PTLD with or without EBV association, confirmed after biopsy or resection
* Measurable disease of > 2 cm in diameter and/or bone marrow involvement
* Patients having undergone heart, lung, liver, kidney, pancreas, small intestine transplantation or other or a combination of the organ transplantations mentioned
* Karnofsky scale >50% or ECOG ≤ 3
* Reduction of immunosuppression with or without antiviral therapy
* A complete surgical extirpation of tumor was not performed
* A radiation therapy was not performed
* Effective contraception for women in childbearing age
* Patient's written informed consent and written consent for data collection
* Patients are > 18 years (or ≥ 15 years with parental agreement )

Exclusion Criteria:

* Life expectancy less than 6 weeks
* Karnofsky-scale <50% or ECOG =3
* Treatment with rituximab before
* Known allergic reactions against foreign proteins
* Concomitant diseases, which exclude the administration of therapy as outlined by the study protocol
* non-compensated heart failure
* Dilatative cardiomyopathy
* Myocardial infarction during the last 6 months
* Severe non-compensated hypertension
* Severe non-compensated diabetes mellitus
* Renal insufficiency (creatinine more than 3-fold of the upper normal value), not related to lymphoma.
* Hepatic insufficiency with transaminase values greater than 3-fold of the normal values and/or bilirubin levels >3.0 mg/dl, not related to lymphoma
* Clinical signs of cerebral dysfunction
* Women during the lactation period, pregnant or of childbearing potential not using a reliable contraceptive method
* Involvement of the central nervous system by the disease
* Severe psychiatric disease
* Known to be HIV positive
* Missing written informed consent of the patient

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2002-12; Primary Completion 2008-05 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
number of patients with complete and partial remission | 1 month (plus or minus 7 days) after the last cycle of chemotherapy
response duration | from date of best response until the date of first documented progression, assessed up to 3 years

SECONDARY OUTCOMES:
number of patients with treatment-related death | from start of treatment, assessed up to 12 months after the end of treatment
overall survival | from start of treatment until date of death from any cause, assessed up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ralf U Trappe, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (4):
- Princess Alexandra Hospital, Ipswich Rd, Woolloongabba, Qld 4102, Brisbane, Australia
- Hôpital Pitié-Salpétrière, Department of Hematology, 47-83 Boulevard de l'Hopital, Paris, France
- Charité - Universitätsmedizin Berlin, Campus Virchow Klinikum, Department of Hematology and Oncology, Augustenburger Platz 1, Berlin, Germany
- Sahlgrens hospital, Department of Hematology, Gothenburg, Sweden

REFERENCES:
- [Derived] Trappe RU, Dierickx D, Zimmermann H, Morschhauser F, Mollee P, Zaucha JM, Dreyling MH, Duhrsen U, Reinke P, Verhoef G, Subklewe M, Huttmann A, Tousseyn T, Salles G, Kliem V, Hauser IA, Tarella C, Van Den Neste E, Gheysens O, Anagnostopoulos I, Leblond V, Riess H, Choquet S. Response to Rituximab Induction Is a Predictive Marker in B-Cell Post-Transplant Lymphoproliferative Disorder and Allows Successful Stratification Into Rituximab or R-CHOP Consolidation in an International, Prospective, Multicenter Phase II Trial. J Clin Oncol. 2017 Feb 10;35(5):536-543. doi: 10.1200/JCO.2016.69.3564. Epub 2016 Dec 19. PMID 27992268
- [Derived] Trappe R, Oertel S, Leblond V, Mollee P, Sender M, Reinke P, Neuhaus R, Lehmkuhl H, Horst HA, Salles G, Morschhauser F, Jaccard A, Lamy T, Leithauser M, Zimmermann H, Anagnostopoulos I, Raphael M, Riess H, Choquet S; German PTLD Study Group; European PTLD Network. Sequential treatment with rituximab followed by CHOP chemotherapy in adult B-cell post-transplant lymphoproliferative disorder (PTLD): the prospective international multicentre phase 2 PTLD-1 trial. Lancet Oncol. 2012 Feb;13(2):196-206. doi: 10.1016/S1470-2045(11)70300-X. Epub 2011 Dec 13. PMID 22173060
- See also: Trial Protocol — http://www.lymphome.de/Gruppen/DPTLDSG/Protokolle/PTLD-I/Protokoll-PTLD-I.pdf